CLINICAL TRIAL: NCT07267871
Title: Oura Blood Pressure Profile Study: An Evaluation of the Oura Blood Pressure Profile Algorithm for Identifying Signs of Hypertension
Brief Title: Oura Blood Pressure Profile Study
Status: Not yet recruiting | Type: Observational
Sponsor: Ouraring Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HTN-2025
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed study is designed as a prospective, single-arm, observational, non-significant risk device study to evaluate the performance of Oura's investigational Blood Pressure Profile algorithm in identifying signs of hypertension.

ELIGIBILITY:
Inclusion Criteria

* Located in United States
* Aged 22 years or older at time of eligibility screener
* Oura Ring user (Oura Ring Gen3 or newer)
* User of the English version of the Oura App
* Smartphone (iOS or Android) user
* Able to provide consent electronically

Exclusion Criteria

* User of implanted cardiac electronic device(s)
* Currently pregnant
* Within 12 weeks postpartum

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include users of the Oura Ring (Gen3 or newer) who are located in the United States and aged 22 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the Oura Blood Pressure Profile classification for identifying participant-reported hypertension | From enrollment until up to 18 months

SECONDARY OUTCOMES:
Specificity of the Oura Blood Pressure Profile classification versus participant-reported hypertension | From enrollment until up to 18 months

OTHER OUTCOMES:
Association between Oura Blood Pressure Profile classification and participant-measured systolic and diastolic blood pressure values | from enrollment until up to 18 months

IPD SHARING:
Plan to Share IPD: Undecided